CLINICAL TRIAL: NCT00917878
Title: The Effects of Milk and Milk Constituents on Postprandial Inflammation in Overweight Subjects
Brief Title: Postprandial Effects of Milk and Milk Constituents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nederlandse Zuivel Organisatie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MEC 08-3-096
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2009-09

CONDITIONS: Hyperlipidemia; Inflammation
Keywords: Milk; Postprandial hyperlipidemia; Postprandial inflammation; Overweight
MeSH Terms: conditions — Hyperlipidemias; Inflammation; Overweight | interventions — Milk; Proteins; Calcium

ARMS (4):
- Milk (Experimental): 500 mL low-fat milk added to high-fat meal
  Interventions: Dietary Supplement: Milk
- Protein (Experimental): Milk protein in 500 mL water added to high-fat meal
  Interventions: Dietary Supplement: Protein
- Calcium (Experimental): Milk calcium in 500 mL water added to high-fat meal
  Interventions: Dietary Supplement: Calcium
- Control (Experimental): Lactose in 500 mL water added to high-fat meal (control condition)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Milk — 500 mL low-fat milk added to high-fat meal
  Arms: Milk
Dietary Supplement: Protein — Milk protein in 500 mL water added to high-fat meal
  Arms: Protein
Dietary Supplement: Calcium — Milk calcium in 500 mL water added to high-fat meal
  Arms: Calcium
Dietary Supplement: Control — Lactose in 500 mL water added to high-fat meal
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether the addition of milk or the milk constituents calcium and protein to a high-fat breakfast affects the postprandial lipid and inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) above 27 kg/m2

Exclusion Criteria:

* Smoking
* Diabetes mellitus
* Cardiovascular diseases
* Familial hypercholesterolemia or lipid lowering medication
* Severe conditions that might interfere with the study outcomes, such as COPD, asthma, rheumatoid arthritis, etc.
* Unstable body weight
* Abuse of alcohol or drugs
* Participation in another biomedical study during the past 30 days
* Having donated blood during the past 30 days

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Plasma inflammatory markers | 6 h after meal

SECONDARY OUTCOMES:
Serum lipids | 6 h after meal

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, Prof. Dr. Ir., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands